CLINICAL TRIAL: NCT05803317
Title: Asymmetry of the Center of Pressure During Gait After Amputation of Lower Limbs
Acronym: ASCOPALL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2023/EP-01
Record Dates: First submitted 2023-03-14; First posted 2023-04-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2024-04

CONDITIONS: Lower Limb Amputation Below Knee (Injury); Lower Limb Amputation Above Knee (Injury)
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amputee patients: All patients with lower limb amputations, unilateral or bilateral, walking with or without technical aids hospitalized in the Rehabilitation Department of the CHU of Nîmes
  Interventions: Other: usual care : Evaluation of walking on a baropodometric platform

INTERVENTIONS:
Other: usual care : Evaluation of walking on a baropodometric platform — Pure observationnal study

SUMMARY:
Retrospective, non-randomized, observational, single-center longitudinal study at the University Rehabilitation Hospital of Grau du Roi CHU of Nîmes, France. From January 2012 to Janvier 2023 patients hospitalized for lower limb amputation, were extracted from the computer database of the motion analysis laboratory (2 baropodometric platforms, Zebris, Germany). All patients with lower limb amputations, unilateral or bilateral, walking with or without technical aids, were included regardless of the level (trans-femoral or trans-tibial). Only patients hospitalized in the locomotor rehabilitation department were included in the study. Patients who were not autonomous for walking and required a third person (human assistance) were not included. Finally, deceased patients were also excluded from the study population. Prior to data collection, all participants received a note of non-objection. The study was reported on the Health Data Hub, and data collection and analysis were performed according to the MR004 reference methodologies.

Walking amputee patients hospitalized in the locomotor rehabilitation department benefited from a systematic gait assessment before discharge from hospital after rehabilitation and validation of the prosthesis. During the gait analysis, on baropodometric platforms, the software provides a number of parameters: spatiotemporal, pressure distribution, vertical component of the ground reaction force and trajectory of the center of pressure. All patients were recorded over a distance of ten meters including the two meters of acceleration and deceleration according to the validity of the TM-10 for a duration of two minutes.

The parameters from the CoP trajectory are calculated from the coordinates calculated in the platform reference frame. A processing of these data will be specially developed within the service. Three key parameters of the COP have been retained: Lateral symmetry (LS; the left/right offset of the intersection point, where the "zero position" is equivalent to perfect symmetry), lateral variability (LV; the standard deviation of the intersection point in the lateral direction, where "zero" equals constant steps in terms of width between the legs), and anteroposterior variability (APV; the standard deviation of the intersection point in the anteroposterior direction, where "zero" equals constant strides while walking on the treadmill). These parameters, which allow for the assessment of continuous COP trajectories with multiple strides, reflect the overall movements of individuals throughout the gait cycle.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral lower limb amputees, walking with or without technical aids, hospitalized in the Locomotor Rehabilitation Department
* Adult patient (≥18 years) and less than 90 years of age.

Exclusion Criteria:

* Patients not autonomous for walking requiring a third person (human assistance) were not included. Finally, deceased patients were also excluded from the study population.
* Patients who objected to the use of their data.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with lower limb amputations, unilateral or bilateral, walking with or without technical aids, whatever the level (trans-femoral or trans-tibial) and hospitalized in the locomotor rehabilitation department of the CHU of Nîmes between January 2012 and January 2023 were included in the study
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Lateral symmetry | Baseline
  Measurement of the lateral symmetry of the center of pressure (LS; the left/right offset of the point of intersection, where the "zero position" is equivalent to perfect symmetry)
Lateral variability | baseline
  Measurement of the Lateral variability of the center of pressure (LV; the standard deviation of the point of intersection in the lateral direction, where "zero" is equivalent to constant steps in terms of width between the legs)
Anteroposterior variability | baseline
  Measurement of the Anteroposterior variability of the center of pressure (APV; the standard deviation of the point of intersection in the anteroposterior direction, where "zero" is equivalent to constant strides while walking on the treadmill)

SECONDARY OUTCOMES:
Walking speed | baseline
  Measurement of the median speed according to the level of amputation and the use or not of a technical aid (in m/sec)

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Pantera E, Reneaud N, Dupeyron A, Pradon D. Impact of amputation level on gait disorders in transfemoral and transtibial amputees. Gait Posture. 2025 Jun;119:23-30. doi: 10.1016/j.gaitpost.2025.02.013. Epub 2025 Feb 21. PMID 40010097